CLINICAL TRIAL: NCT06744322
Title: Fast Discharge After Acute Myocardial Infarction Discharge MI - A Randomized Multicenter Non Inferiority Trial
Brief Title: Fast Discharge After Acute Myocardial Infarction Discharge MI
Acronym: DISCHARGE-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1284/2024; 20241113-3609 (Other: Medical University Innsbruck)
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-11

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Myocardial Infarction; STEMI; NSTEMI; Discharge; Randomized
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention): Patients undergo a standard post-infarction care, with discharge at 72 (+/-24 hours) after invasive management of acute myocardial infarction.
- Fast discharge strategy (Experimental): Fast discharge at 24 (+/-12) hours after invasive management of acute myocardial infarction.
  Interventions: Procedure: Fast discharge strategy

INTERVENTIONS:
Procedure: Fast discharge strategy — Patients undergoing invasive management after myocardial infarction will be discharged after 24 (+/- 12) hours.
  Arms: Fast discharge strategy

SUMMARY:
To evaluate the hypothesis that a fast discharge strategy (discharge at 24 [± 12] hours) following invasive management for acute myocardial infarction is non-inferior to standard of care (72 [± 24] hours) with respect to the risk of major adverse cardiovascular events (MACE) at 12 months.

DETAILED DESCRIPTION:
The goal of this randomized, multicenter trial is to assess the safety of a fast discharge strategy following acute myocardial infarction as compared to standard of care. The trial will evaluate the hypothesis that a fast discharge strategy (discharge at 24 [± 12] hours) following invasive management of acute myocardial infarction is non-inferior to standard of care (discharge at 72 [± 24] hours) with respect to the risk of major adverse cardiovascular events at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated acute myocardial infarction (NSTEMI and STEMI) diagnosed according to the 2023 acute coronary syndrome guidelines of the ESC
* Age ≥ 18 years at time of consent
* Invasive management strategy and in case of PCI successful intervention of the culprit lesion defined by post-interventional TIMI 3 flow
* Absence of PCI-related complications (coronary perforation, side branch closure, inability to deliver stent/balloon, aortic dissection, allergic reaction grade ≥2, stroke/thromboembolism, access site complications including pseudoaneurysm, arteriovenous fistula, retroperitoneal hemorrhage and arterial dissection/occlusion or emboli)
* Ability to understand and willingness to sign and date written informed consent

Exclusion Criteria:

* Myocardial infarction complicated by cardiac arrest (out-of-hospital cardiac arrest/in-hospital cardiac arrest)
* Malignant arrhythmias including sustained ventricular arrhythmias and persistent bradycardia (< 50 beats per minute due to sinus node or atrioventricular conduction system abnormalities, second- /third-degree atrioventricular block) after PCI
* Ongoing hemodynamic instability (systolic blood pressure <90 mmHg, elevated lactate concentrations, need for inotropes or vasopressors)
* Ongoing respiratory instability defined by Killip class >I (rales, pulmonary edema)
* Ongoing quantitative disorders of consciousness (somnolence, sopor, coma)
* Pregnancy
* Immobility/limited mobility or social circumstances that prevent fast discharge assessed by an interprofessional care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2224 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | At 12 months
  MACE is defined as a composite of all-cause death, myocardial re-infarction and unscheduled cardiovascular re-hospitalization.

SECONDARY OUTCOMES:
All cause death | At 30 days at 12 months
  Death from any cause.
Myocardial re-infarction | At 30 days and 12 months
  Number of patients experiencing myocardial re-infarction
Unscheduled cardiovascular re-hospitalization | At 30 and12 months
  Unscheduled cardiovascular re-hospitalization
Cardiovascular death | At 30 days and 12 months
  Number of patients experiencing cardiovascular-related death
Heart failure hospitalization | At 30 days and 12 months
  Number of patients hospitalized for heart failure
Stroke | At 30 days and 12 months
  Number of patients experiencing a stroke
Bleeding events | At 30 days and 12 months
  Number of bleeding events at 12 months
Cost-effectiveness | At 12 months
  Cost-effectiveness measurements
Length of hospital stay | Hospitalization
  Number of days in hospital from time of infarction to hospital discharge
Percentage of patients on guideline-directed therapy | At 30 days and 12 months.
  Percentage of patients on guideline-directed therapy

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reindl, MD, PhD, Principal Investigator — Medical University Innsbruck; Sebastian J Reinstadler, MD, PhD, Principal Investigator — Medical University of Innsbruck
Locations (8):
- Austria (7):
  - Hospital Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg, Salzburg, Salzburg
  - Cardinal Schwarzenberg Hospital Schwarzach, Schwarzach im Pongau, Schwarzach Im Pongau
  - Medical University of Graz, Graz, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - University Teaching Hospital Wels-Grieskirchen, Wels, Upper Austria
  - Academic Teaching Hospital Feldkirch, Feldkirch, Vorarlberg
- Ludwig Maximilian University Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No